CLINICAL TRIAL: NCT03298997
Title: Comparison Between the Ligation and Hemorrhoidopexy Technique and the Conventional Ligation of Hemorrhoidal Arteries Using Ultrasound: a Prospective, Randomized Controlled Study
Brief Title: Ligation and Hemorrhoidopexy Technique Versus Ligation of Hemorrhoidal Arteries Using Ultrasound for Hemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Perivoliotis Konstantinos, Perivoliotis Konstantinos MD, MSc Principal Investigator, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hemorrhoids RCT
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Ligation; Ultrasound; Prospective; Randomized Controlled Trial
MeSH Terms: conditions — Hemorrhoids | interventions — Ligation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding will exist at the level of the patient and the investigator who will record the data postoperatively, regarding the surgical technique applied. There will be no blinding at the level of the surgeon and the anesthesiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligation and Hemorrhoidopexy (Experimental): The patient will be placed in the Lloyd-Davies position. Provision of a sterile field, using a 10% povidone iodine solution. Rectal dilatation will be performed with a 10% xylocaine gel. Introduction of a proctoscope. Identification of the hemorrhoidal nodules (3rd, 7th, 11th hour). Confirmation of the hemorrhoidal artery location, through palpation. Ligation of the hemorrhoidal nodules using an absorbable polyglycolic acid suture (2-0, 5/8 inch needle).
  Placement of a fixative suture in the hemorrhoidal nodule and then performance of hemorrhoidopexy Placement of a hemostatic gauze in the surgical field. Prior to operation, the patients will be submitted to pudendal nerve block. Using an atraumatic 25 Gauge (G) needle, a 20ml lidocaine solution (diluted with saline in a 1:1 rate) will be administered bilaterally, medially to the ischial tuberosity.
  10 minutes before the operation, the patient will receive 1-2.5mg midazolam and 0.1-0.2 mg fentanyl.
  Interventions: Procedure: Ligation and Hemorrhoidopexy
- Ultrasound Guided Ligation of Hemorrhoidal Arteries (Active Comparator): The patient will be placed in the Lloyd-Davies position. Provision of a sterile field, using a 10% povidone iodine solution. Rectal dilatation will be performed with a 10% xylocaine gel. Use of a proctoscope combined with a Doppler sensor. After the hemorrhoidal artery localization, Z ligations will be placed, using an absorbable polyglycolic acid suture (2-0, 5/8 inch needle).
  The proper artery ligation will be confirmed by the absence of the Doppler signal.
  In the presence of residual hemorrhoidal tissue hemorrhoidopexy will be performed, by applying a continuous suture.
  Placement of a hemostatic gauze in the surgical field. Prior to operation, the patients will be submitted to spinal anesthesia. Using an atraumatic 25 Gauge (G) needle, a levobupivacaine 5mg/ml and fentanyl 25mg solution, will be administered at the height of lumbar (L)2-L3 or L3-L4.
  Interventions: Procedure: Ultrasound Guided Ligation of Hemorrhoidal Arteries

INTERVENTIONS:
Procedure: Ligation and Hemorrhoidopexy — Identification through palpation and ligation of the hemorrhoidal nodules (3rd, 7th, 11th hour), using an absorbable polyglycolic acid suture (2-0, 5/8 inch needle).
  Prior to operation, the patients will be submitted to pudendal nerve block.
  Arms: Ligation and Hemorrhoidopexy
Procedure: Ultrasound Guided Ligation of Hemorrhoidal Arteries — Ultrasound guided identification and ligation of the hemorrhoidal arteries, using an absorbable polyglycolic acid suture (2-0, 5/8 inch needle).
  Prior to operation, the patients will be submitted to spinal anesthesia.
  Arms: Ultrasound Guided Ligation of Hemorrhoidal Arteries

SUMMARY:
The purpose of this study is to compare two techniques for treating hemorrhoids, the ligation and hemorrhoidopexy technique and the conventional ligation of hemorrhoidal arteries using ultrasound, in patients with non-complicated hemorrhoids.

DETAILED DESCRIPTION:
Surgical operations for the treatment of perianal diseases are a major part of all elective surgical cases. The reduction in the hospitalization time of patients undergoing surgical procedures for benign perianal diseases is to the benefit of both the patient and healthcare provider. The importance of 'one day' surgical operations lies in the fact that the patient returns directly to his social and working environment, while the number of occupied hospital beds and the total hospitalization costs are reduced. A typical example is the goal set by National Health Service (NHS), where the 75% of the scheduled operations should consist of 'one day' operations. In order to achieve this goal, several obstacles should be dealt with, including the implementation of more efficient and safe surgical techniques. Therefore, this would be associated with a decrease in the operation time, early recovery and faster hospital discharge.

Hemorrhoids is one of the most common benign perianal diseases. According to a recent prospective study of 976 patients, 38.93% of them suffered from hemorrhoids, with 8.16% and 0.53% being Grade III and IV, according to Goligher classification, respectively. The percentage of the symptomatic patients was, also, significant (44.74%). Symptomatic hemorrhoids, include bleeding, pruritus, pain, poor hygiene and the presence of palpable hemorrhoid nodules.

As far as the blood supply of the rectum and the broader anatomic region is concerned, it is provided by the superior, middle and inferior hemorrhoidal arteries. The superior hemorrhoidal artery is a branch of the inferior mesenteric artery and is carried behind the rectum, where it provides branches up to the internal sphincter muscle. The right and left middle hemorrhoidal artery originate from the respective internal iliac artery and their branches are cross-linked with the respective branches deriving from the superior hemorrhoidal artery. Finally, inferior hemorrhoidal arteries derive from the respective internal pudendal arteries. Correspondingly, hemorrhoidal venous plexus consists of the middle and inferior hemorrhoidal veins, which through the internal iliac veins drain into the inferior cava vein. Hemorrhoidal tissue constitutes a continence mechanism of the upper rectum and consists of vascular tissue, connective tissue and smooth muscle fibers, within the rectal canal. Through the approximation of the hemorrhoidal tissue, closure of the anal canal and protection of the sphincter mechanism is achieved. Since modern pathogenesis theories of hemorrhoidal disease attribute to the increased arterial flow in the hemorrhoidal plexus the generating cause of this disease, recent anatomical studies mapped the vascular network, indicating that the arteries are not confined to the anatomical regions described in the literature.

According to recent guidelines, the modification of dietary intake, through the increase of fluid and fiber intake, consists the first line treatment of symptomatic hemorrhoidal disease. However, in Grade III-IV hemorrhoidal disease or in Grade II, where conservative therapy failed, surgical intervention is required. Surgeon has plenty of techniques at his disposal, in order to treat hemorrhoids. Examples of these techniques are operations, such as hemorrhoidectomy (open, closed, Milligan-Morgan, Parks, using staplers, using energy sources, e.g. Harmonic, Ligasure, Laser, bipolar forceps), elastic rings ligation, sclerotherapy and Hemorrhoidal Arteries Ligation (ΗΑL) or Transanal Hemorrhoidal Dearterialization (THD).

Ligation of hemorrhoidal arteries using a Doppler apparatus, is a minimally invasive technique that was first applied by Morinaga et al. in 1995 and has as principle the elective ligation of the arteries that supply the hemorrhoidal plexus. In a recent meta-analysis, the superiority of HAL in areas such as, postoperative bleeding, emergency reoperation, operative duration, length of hospital stay and postoperative pain, was shown. A major drawback of this technique, however, remains the high rate of recurrence, which ranges from 11.1% to 59.3%, for Grade IV hemorrhoids.

Despite the comparative advantages of this minimally invasive technique, the high cost of the necessary equipment and the respective consumables, is a barrier to its broad application. Gupta et al. in a prospective randomized study, compared Doppler-Guided HAL (DG-HAL) to hemorrhoid artery ligation and hemorrhoidopexy. Ligation was performed on the hemorrhoid nodule at the 3rd, 7th and 11th hours, followed by continuous hemorrhoidal nodule ligation and hemorrhoidopexy. The DG-HAL group had a significantly longer operative time (31 min vs 9 min) and post-operative pain (4.4 vs 2.2), without any differences in complication or recurrence rates. Similarly, Huang et al., reported a respective ligation technique, where, through the use of the index finger, the artery was palpated, followed by repeating compression and ligation cycles, in order to fix the affected hemorrhoids above the dental line. In this group, operative time was longer when compared to the DG-HAL group (35.57 vs. 12.73). There was no difference in terms of postoperative improvement of symptoms and hospitalization duration. In the experimental group, however, the cost of hospitalization and the relapse rate was significantly lower. Finally, Aigner et al., in a recent randomized study, investigated the efficacy of hemorrhoidopexy for Grade III hemorrhoids. They concluded that the techniques of hemorrhoidopexy are effective and the addition of DG-HAL does not affect the results.

Given these facts, the present trial was designed, in order to compare the two techniques for hemorrhoidal disease treatment, the ligation and hemorrhoidopexy technique and the conventional ligation of hemorrhoid arteries using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Μale or female
* Age: 18 to 80 years
* American Society of Anesthesiologists (ASA) score: I and II
* Grade I, II, and III hemorrhoids

Exclusion Criteria:

* Acute perianal diseases, such as perianal abscesses, complicated hemorrhoids (e.g., thrombosis) and acute anal fissure
* Malignant perianal disorders
* Patient age ≥ 80 years
* ASA score ≥ ΙΙΙ
* Presence of inflammatory bowel disease
* History of a previous rectoanal operation
* Presence of a clinically significant cardiovascular, respiratory, renal, hepatic or metabolic disorder. Furthermore, diseases, such as obesity, psychiatric disorders or gastrointestinal disorders constitute exclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Symptoms Remission Rate | 1 month postoperatively
  The primary endpoint of the present study, is the identification of difference in the symptoms remission rate, within one month postoperatively, between the ligation and hemorrhoidopexy technique and the conventional ligation of hemorrhoidal arteries using ultrasound, in patients with non-complicated hemorrhoidal disease.
  If the symptoms are treated then it will be defined as=1 'YES' If the symptoms are not treated then it will be defined as=0 'NO'

SECONDARY OUTCOMES:
Operative time | Intraoperative period
  The total operative time will be recorded. Measurement unit: minutes
Postoperative mobilization time | Maximum time frame 24 hours postoperatively
  The postoperative mobilization time of the patient will be recorded. Measurement unit: hours
Onset of oral feeding | Maximum time frame 24 hours postoperatively
  The time that the patient started oral feeding will be recorded. Measurement unit: hours
Postoperative pain level at 12 hours | 12 hours postoperatively
  Postoperative pain level at 12 hours after surgery, quantified with the use of the Visual analogue scale (VAS) scale.
Hypotension | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative hypotension. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Nausea | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative nausea. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Vomiting | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative vomiting. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Headache | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative headache. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Urinary retention | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative urinary retention. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Bleeding at the operative site | Maximum time frame 24 hours postoperatively
  Occurrence of postoperative bleeding at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Postoperative discharge time | Maximum time frame 48 hours postoperatively
  Postoperative time that the patient can be safely discharged. Measurement unit: hours.
  The patient will be discharged, when it is ensured that is medically safe to be released. In particular, as the exit time of the patient, will be regarded the time that the patient will fulfill the Clinical Discharge Criteria. More specifically, the patient should meet the following : steady vital signs, be oriented, without nausea or vomiting, mobilized with a steady gait, without a significant bleeding.
Postoperative pain level at 7 days | 7 days postoperatively
  Postoperative pain level at 7 days after surgery, quantified with the use of the VAS scale.
Oedema at the operative site | 7 days postoperatively
  Occurrence of postoperative oedema at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Hematoma at the operative site | 7 days postoperatively
  Occurrence of postoperative hematoma at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Infection at the operative site | 7 days postoperatively
  Occurrence of postoperative infection at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Stenosis at the operative site | 7 days postoperatively
  Occurrence of postoperative stenosis at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Postoperative return to work time | Postoperative period up to 1 month
  The time that the patient resumed his work or normal activities will be recorded. Measurement unit: days
Pruritus | 1 year postoperatively
  Occurrence of postoperative pruritus at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Mucosal proptosis | 1 year postoperatively
  Occurrence of postoperative mucosal proptosis at the operative site. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Perianal nodules | 1 year postoperatively
  Occurrence of postoperative perianal nodules. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Constipation | 1 year postoperatively
  Occurrence of postoperative constipation. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Tenesmus | 1 year postoperatively
  Occurrence of tenesmus. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Reoperation | 1 year postoperatively
  Occurrence of reoperation. If the patient is reoperated, then it will be defined as=1 'YES' If the patient is not reoperated, then it will be defined as=0 'NO'
Disease recurrence rate | 1 year postoperatively
  Disease recurrence rate If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Satisfaction level | 1 year postoperatively
  Satisfaction level measured at a 0-10 scale
Difference in the quality of life of the patient | Preoperatively, 1 month postoperatively and 1 year postoperatively
  Difference in the quality of life of the patient, at 1 month and 1 year postoperatively, compared to the respective preoperative measurements, based on the Short Form 36 (SF-36) questionnaire, weighted for the Greek population.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tepetes, Professor, Study Director — Department of Surgery, University Hospital of Larissa
Locations (1):
- Department of Surgery, University Hospital of Larissa, Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faiz OD, Brown TJ, Colucci G, Grover M, Clark SK. Trends in colorectal day case surgery in NHS Trusts between 1998 and 2005. Colorectal Dis. 2008 Nov;10(9):935-42. doi: 10.1111/j.1463-1318.2008.01481.x. Epub 2008 Feb 21. PMID 18294271
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Schuurman JP, Go PM, Bleys RL. Anatomical branches of the superior rectal artery in the distal rectum. Colorectal Dis. 2009 Nov;11(9):967-71. doi: 10.1111/j.1463-1318.2008.01729.x. Epub 2008 Oct 31. PMID 19175645
- [Background] Rivadeneira DE, Steele SR, Ternent C, Chalasani S, Buie WD, Rafferty JL; Standards Practice Task Force of The American Society of Colon and Rectal Surgeons. Practice parameters for the management of hemorrhoids (revised 2010). Dis Colon Rectum. 2011 Sep;54(9):1059-64. doi: 10.1097/DCR.0b013e318225513d. No abstract available. PMID 21825884
- [Background] Ho YH, Seow-Choen F, Tan M, Leong AF. Randomized controlled trial of open and closed haemorrhoidectomy. Br J Surg. 1997 Dec;84(12):1729-30. PMID 9448627
- [Background] Hosch SB, Knoefel WT, Pichlmeier U, Schulze V, Busch C, Gawad KA, Broelsch CE, Izbicki JR. Surgical treatment of piles: prospective, randomized study of Parks vs. Milligan-Morgan hemorrhoidectomy. Dis Colon Rectum. 1998 Feb;41(2):159-64. doi: 10.1007/BF02238242. PMID 9556238
- [Background] Senagore AJ, Singer M, Abcarian H, Fleshman J, Corman M, Wexner S, Nivatvongs S; Procedure for Prolapse and Hemmorrhoids (PPH) Multicenter Study Group. A prospective, randomized, controlled multicenter trial comparing stapled hemorrhoidopexy and Ferguson hemorrhoidectomy: perioperative and one-year results. Dis Colon Rectum. 2004 Nov;47(11):1824-36. doi: 10.1007/s10350-004-0694-9. PMID 15622574
- [Background] Chung CC, Cheung HY, Chan ES, Kwok SY, Li MK. Stapled hemorrhoidopexy vs. Harmonic Scalpel hemorrhoidectomy: a randomized trial. Dis Colon Rectum. 2005 Jun;48(6):1213-9. doi: 10.1007/s10350-004-0918-z. PMID 15793648
- [Background] Lawes DA, Palazzo FF, Francis DL, Clifton MA. One year follow up of a randomized trial comparing Ligasure with open haemorrhoidectomy. Colorectal Dis. 2004 Jul;6(4):233-5. doi: 10.1111/j.1463-1318.2004.00608.x. PMID 15206964
- [Background] Pandini LC, Nahas SC, Nahas CS, Marques CF, Sobrado CW, Kiss DR. Surgical treatment of haemorrhoidal disease with CO2 laser and Milligan-Morgan cold scalpel technique. Colorectal Dis. 2006 Sep;8(7):592-5. doi: 10.1111/j.1463-1318.2006.01023.x. PMID 16919112
- [Background] Chung CC, Ha JP, Tai YP, Tsang WW, Li MK. Double-blind, randomized trial comparing Harmonic Scalpel hemorrhoidectomy, bipolar scissors hemorrhoidectomy, and scissors excision: ligation technique. Dis Colon Rectum. 2002 Jun;45(6):789-94. doi: 10.1007/s10350-004-6299-5. PMID 12072632
- [Background] Shanmugam V, Thaha MA, Rabindranath KS, Campbell KL, Steele RJ, Loudon MA. Systematic review of randomized trials comparing rubber band ligation with excisional haemorrhoidectomy. Br J Surg. 2005 Dec;92(12):1481-7. doi: 10.1002/bjs.5185. PMID 16252313
- [Background] Khoury GA, Lake SP, Lewis MC, Lewis AA. A randomized trial to compare single with multiple phenol injection treatment for haemorrhoids. Br J Surg. 1985 Sep;72(9):741-2. doi: 10.1002/bjs.1800720924. PMID 3899248
- [Background] Ratto C, Donisi L, Parello A, Litta F, Doglietto GB. Evaluation of transanal hemorrhoidal dearterialization as a minimally invasive therapeutic approach to hemorrhoids. Dis Colon Rectum. 2010 May;53(5):803-11. doi: 10.1007/DCR.0b013e3181cdafa7. PMID 20389215
- [Background] Morinaga K, Hasuda K, Ikeda T. A novel therapy for internal hemorrhoids: ligation of the hemorrhoidal artery with a newly devised instrument (Moricorn) in conjunction with a Doppler flowmeter. Am J Gastroenterol. 1995 Apr;90(4):610-3. PMID 7717320
- [Background] Simillis C, Thoukididou SN, Slesser AA, Rasheed S, Tan E, Tekkis PP. Systematic review and network meta-analysis comparing clinical outcomes and effectiveness of surgical treatments for haemorrhoids. Br J Surg. 2015 Dec;102(13):1603-18. doi: 10.1002/bjs.9913. Epub 2015 Sep 30. PMID 26420725
- [Background] Giordano P, Overton J, Madeddu F, Zaman S, Gravante G. Transanal hemorrhoidal dearterialization: a systematic review. Dis Colon Rectum. 2009 Sep;52(9):1665-71. doi: 10.1007/DCR.0b013e3181af50f4. PMID 19690499
- [Background] Gupta PJ, Kalaskar S, Taori S, Heda PS. Doppler-guided hemorrhoidal artery ligation does not offer any advantage over suture ligation of grade 3 symptomatic hemorrhoids. Tech Coloproctol. 2011 Dec;15(4):439-44. doi: 10.1007/s10151-011-0780-7. Epub 2011 Oct 28. PMID 22033542
- [Background] Gupta PJ, Kalaskar S. Ligation and mucopexy for prolapsing hemorrhoids--a ten year experience. Ann Surg Innov Res. 2008 Nov 28;2:5. doi: 10.1186/1750-1164-2-5. PMID 19038061
- [Background] Huang HX, Yao YB, Tang Y. Application of 'tying, binding and fixing operation' in surgical treatment of severe mixed hemorrhoids. Exp Ther Med. 2016 Aug;12(2):1022-1028. doi: 10.3892/etm.2016.3339. Epub 2016 May 12. PMID 27446315
- [Background] Aigner F, Kronberger I, Oberwalder M, Loizides A, Ulmer H, Gruber L, Pratschke J, Peer S, Gruber H. Doppler-guided haemorrhoidal artery ligation with suture mucopexy compared with suture mucopexy alone for the treatment of Grade III haemorrhoids: a prospective randomized controlled trial. Colorectal Dis. 2016 Jul;18(7):710-6. doi: 10.1111/codi.13280. PMID 26787597
- [Background] Spyridakis M, Christodoulidis G, Symeonidis D, Dimas D, Diamantis A, Polychronopoulou E, Tepetes K. Outcomes of Doppler-guided hemorrhoid artery ligation: analysis of 90 consecutive patients. Tech Coloproctol. 2011 Oct;15 Suppl 1:S21-4. doi: 10.1007/s10151-011-0727-z. PMID 21887577
- [Background] Tepetes K, Symeonidis D, Christodoulidis G, Spyridakis M, Hatzitheofilou K. Pudendal nerve block versus local anesthesia for harmonic scalpel hemorrhoidectomy: a prospective randomized study. Tech Coloproctol. 2010 Nov;14 Suppl 1:S1-3. doi: 10.1007/s10151-010-0614-z. PMID 20683750
- [Background] Honca M, Dereli N, Kose EA, Honca T, Kutuk S, Unal SS, Horasanli E. Low-dose levobupivacaine plus fentanyl combination for spinal anesthesia in anorectal surgery. Braz J Anesthesiol. 2015 Nov-Dec;65(6):461-5. doi: 10.1016/j.bjane.2014.01.007. Epub 2014 Feb 20. PMID 26614142
- [Background] Alkhaldi HM, Salaita WM, Shabaneh MA, Al-Horut MI, Aldabbas RM, Uraiqat AA. Postoperative Outcome Comparison Between Pudendal Nerve Block and Caudal Block After Lateral Open Internal Sphincterotomy. Med Arch. 2015 Jun;69(3):187-9. doi: 10.5455/medarh.2015.69.187-189. Epub 2015 Jun 10. PMID 26261389
- [Background] Pappa E, Kontodimopoulos N, Niakas D. Validating and norming of the Greek SF-36 Health Survey. Qual Life Res. 2005 Jun;14(5):1433-8. doi: 10.1007/s11136-004-6014-y. PMID 16047519
- [Background] Flight L, Julious SA. Practical guide to sample size calculations: non-inferiority and equivalence trials. Pharm Stat. 2016 Jan-Feb;15(1):80-9. doi: 10.1002/pst.1716. Epub 2015 Nov 25. PMID 26604186
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Result] Perivoliotis K, Spyridakis M, Zintzaras E, Arnaoutoglou E, Pramateftakis MG, Tepetes K. An enhanced outpatient modality for the treatment of hemorrhoidal disease: preliminary results. G Chir. 2019 Mar-Apr;40(2):153-157. PMID 31131818
- [Result] Perivoliotis K, Spyridakis M, Zintzaras E, Arnaoutoglou E, Pramateftakis MG, Tepetes K. Non-Doppler hemorrhoidal artery ligation and hemorrhoidopexy combined with pudendal nerve block for the treatment of hemorrhoidal disease: a non-inferiority randomized controlled trial. Int J Colorectal Dis. 2021 Feb;36(2):353-363. doi: 10.1007/s00384-020-03768-8. Epub 2020 Oct 6. PMID 33025104

DOCUMENTS (3):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03298997/Prot_002.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03298997/ICF_003.pdf
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03298997/SAP_004.pdf